CLINICAL TRIAL: NCT03732326
Title: Effects of Bariatric Surgery on Cardiac and Vascular Structure and Function in Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, The chief director of department of cardiology, Shanghai 10th People's Hospital
Other Study IDs: B-VAS
Record Dates: First submitted 2018-11-01; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Bariatric Surgery
Keywords: Cardiac and Vascular Structure and Function
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bariatric surgery — Bariatric surgery for enrolled patients who fulfill the including criteria

SUMMARY:
This is a prospective cohort study which aims to explore the effect of bariatric surgery on cardiac and vascular structure and function in obesity. Enrolled patients will receive the following examinations before surgery and 3,6,12 month after the bariatric surgery: 24-h central and brachial ambulatory blood pressure monitoring, PWV, echocardiography, vascular endothelial function, hemodynamic including cardiac output and peripheral vascular resistance and so on. We compare these data before and after surgery in order to evaluate effectiveness of bariatric surgery in the cardiac and vascular structure and function.

DETAILED DESCRIPTION:
The including citeria: 1)15-65 years old; 2) Indication for Asian bariatric surgery (I.BMI≥32.5 or 27.5≤BMI<32.5 with obesity-related comorbidities ) ;3) available for inspection and therapeutic schedule; 4) available for follow up. The excluding cteria: 1)over 65 years old; 2)myocardial infarction, angina pectoris and ischemic stroke during the previous month;3)congestive heart failure class IV based on the New York Heart Association classification; 4) malignancy or any other condition with poor prognosis; 5) serious pulmonary and renal dysfunction; 6) gastric disease; 7) poor compliance 8) incomplete clinical data .After enrollment, every patient will receive a question-based interview to obtain medical history and the following examinations and tests: anthropometric parameters measurement including body height, weight, waist circumference, hip circumference and so on; blood routine tests and biochemical tests. Every patient needs to be assessed before surgery and at 3,6,12 month by 24-h central and brachial ambulatory blood pressure, PWV, echocardiography, vascular endothelial function, cardiac output and peripheral vascular resistance. We compare these data before and after surgery in order to evaluate effectiveness of bariatric surgery in the vascular structure and function.

ELIGIBILITY:
Inclusion Criteria:

* 15-65 years old
* conformed indication of Asian bariatric surgery (I.BMI≥32.5 or 27.5≤BMI<32.5 with obesity-related comorbidities )
* available for inspection and therapeutic schedule
* available for follow up

Exclusion Criteria:

* over 65 years old
* myocardial infarction, angina pectoris and ischemic stroke during the previous month
* congestive heart failure class IV based on the New York Heart Association classification
* malignancy or any other condition with poor prognosis
* serious pulmonary and renal dysfunction
* gastric disease
* poor compliance
* incomplete clinical data

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with morbid obesity, aged 15-65 years and without other severe diseases such as congestive heart failure, serious pulmonary and renal dysfunction and so forth.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-01-24 (Estimated); Study Completion 2019-10-24 (Estimated)

PRIMARY OUTCOMES:
left ventricular mass index | 1 year
  changes of left ventricular mass index representing cardiac structure measured by ultrasound will be seen from baseline at 1 year
value of E and A peak | 1 year
  changes of value of E and A peak representing cardiac diastolic function measured by ultrasound will be seen from baseline at 1 year
EF | 1 year
  changes of EF representing cardiac systolic function measured by ultrasound will be seen from baseline at 1 year
pulse wave velocity | 1 year
  changes of pulse wave velocity representing vascular structure measured by SphygmoCor will be seen from baseline at 1 year
flow-mediated dilatation | 1 year
  changes of flow-mediated dilatation representing vascular function measured by UNEX EF will be seen from baseline at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, MD, PhD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taegtmeyer H, Leichman JG, Reyes M, Lux TR. Early benefits from weight-loss surgery. J Am Coll Cardiol. 2010 Apr 20;55(16):1754; author reply 1754. doi: 10.1016/j.jacc.2009.11.081. No abstract available. PMID 20394883
- [Result] Rider OJ, Francis JM, Ali MK, Petersen SE, Robinson M, Robson MD, Byrne JP, Clarke K, Neubauer S. Beneficial cardiovascular effects of bariatric surgical and dietary weight loss in obesity. J Am Coll Cardiol. 2009 Aug 18;54(8):718-26. doi: 10.1016/j.jacc.2009.02.086. PMID 19679250
- [Result] Petersen KS, Clifton PM, Lister N, Keogh JB. Effect of weight loss induced by energy restriction on measures of arterial compliance: A systematic review and meta-analysis. Atherosclerosis. 2016 Apr;247:7-20. doi: 10.1016/j.atherosclerosis.2016.01.042. Epub 2016 Jan 29. PMID 26854971